CLINICAL TRIAL: NCT05312151
Title: The Safety and Tolerability of COMP360 in Participants With Post-traumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: COMPASS Pathways (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMP 201
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: psilocybin; COMP360; COMPASS; PTSD; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- COMP360 Psilocybin (Experimental): 25 mg COMP360 Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Open label
  Other Names: COMP360

SUMMARY:
The Safety and Tolerability of COMP360 in Participants with Post-traumatic Stress Disorder

DETAILED DESCRIPTION:
The Safety and Tolerability of COMP360 administered under supportive conditions in participants with Post-traumatic Stress Disorder

ELIGIBILITY:
Key Inclusion Criteria:

* Meet DSM-5 criteria for current PTSD resulting from a trauma experienced during adulthood measured via the PCL-5 in combination with the LEC-5 at screening
* Meet DSM-5 criteria for current PTSD resulting from a trauma experienced during adulthood as assessed by the CAPS, with a minimum score of 25 at baseline
* Able to identify a next of kin who is willing and able to be reached by the investigators in case of emergency
* Have successfully discontinued all prohibited medications at least two weeks prior to baseline visit. For fluoxetine (Prozac), immediate cessation at screening period visit 1a followed by at least four weeks of run-in will be required prior to baseline

Key Exclusion Criteria:

* Current or past history of schizophrenia, schizoaffective disorder or any other form of psychotic disorder, obsessive compulsive disorder, personality disorders, bipolar disorder, or any other significant disorder as assessed by clinician judgement and a structured clinical interview (MINI 7.0.2)
* Diagnosis of complex PTSD according to clinician judgement
* Borderline Personality Disorder as demonstrated by both the McLean Screening Instrument for Borderline Personality Disorder (MSI- BPD) score ≥ 7 and clinical confirmation of diagnosis by the study clinician and Medical Monitor
* Significant suicide risk as defined by (1) suicidal ideation as endorsed on items 4 or 5 on the C-SSRS within the past year, during screening or at baseline, or; (2) suicidal behaviours within the past year, or; (3) history of serious suicide attempt that required a rescuing medical intervention, or; (4) clinical assessment of significant suicidal risk during participant interview
* Current (within the last year) alcohol or substance use disorder as informed by DSM-5 assessed via the MINI 7.0.2 at screening
* Other personal circumstances and behaviour judged to be incompatible with establishment of rapport or safe exposure to psilocybin
* Exposure to 3,4-methylenedioxymethamphetamine (MDMA), psilocybin, or any other psychedelics, such as ayahuasca, mescaline, lysergic acid diethylamide (LSD), or peyote in the past year
* Primary diagnosis of major depressive disorder within 6 months of study entry
* Exposure to a traumatic experience in the past 3 months
* Significant childhood physical or sexual abuse based on clinician judgment with the use of CTQ
* Enrolment in a psychological therapy programme that will not remain stable for the duration of the study. Psychological therapies cannot have been initiated within 21 days of baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Sunstone Therapies, Rockville, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
- Kings College London, Institute of Psychiatry, Psychology and Neurology, London, United Kingdom

REFERENCES:
- [Derived] Modlin NL, Williamson V, Goodwin GM, Malievskaia E, Atli M, Elek Z, Gaillard A, Koelpin D, Cleare A, Agrawal M, Yehuda R, Kirlic N, Rucker J. Investigational psilocybin treatment for post-traumatic stress disorder: a qualitative study of participant experience, trauma engagement, and differences from standard treatment. EClinicalMedicine. 2025 Dec 5;90:103692. doi: 10.1016/j.eclinm.2025.103692. eCollection 2025 Dec. PMID 41497513
- [Derived] McGowan NM, Rucker JJ, Yehuda R, Agrawal M, Modlin NL, Simmons H, Tofil-Kaluza A, Das S, Goodwin GM. Investigating the safety and tolerability of single-dose psilocybin for post-traumatic stress disorder: A nonrandomized open-label clinical trial. J Psychopharmacol. 2025 Aug 29:2698811251362390. doi: 10.1177/02698811251362390. Online ahead of print. PMID 40883964

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COMP360 Psilocybin
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set - all participants who received study drug.
Arm/Group | COMP360 Psilocybin
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
  United Kingdom | 13
CAPS-5 Total Symptom Severity Score [Mean (Standard Deviation); unit: units on a scale] | 47.5 (9.78)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: A TEAE is defined as an adverse event (AE) that has an onset on or after the dose of study drug, or any pre-existing AE condition that has worsened on or after the dose of study drug.
Time Frame: Up to 12 weeks
Population: Safety Analysis Set - all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | COMP360 Psilocybin
Number analyzed (Participants) | 22
Participants | 22

2. Secondary Outcome: Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Severity Score From Baseline
Description: CAPS-5 is a 30 item scale, each item is scored from 0-4, total severity score is calculated by taking the sum of the individual item scores (range: 0-80). Higher scores denote greater symptom severity.
Time Frame: Week 12
Population: Full Analysis Set - all participant who received study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COMP360 Psilocybin
Number analyzed (Participants) | 22
units on a scale | -29.5 (15.43)

3. Secondary Outcome: Proportion of Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Responders
Description: CAPS-5 is a 30 item scale, each item is scored from 0-4, total severity score is calculated by taking the sum of the individual item scores (range: 0-80). Higher scores denote greater symptom severity.
  A participant is defined as a responder if they have a greater than or equal to 15 point improvement on the CAPS-5 total severity score compared to Baseline.
Time Frame: Week 12
Population: Full Analysis Set - all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | COMP360 Psilocybin
Number analyzed (Participants) | 22
Participants | 17

4. Secondary Outcome: Proportion of Clinician-Administered PTSD Scale From DSM-5 (CAPS-5) Remitters.
Description: CAPS-5 is a 30 item scale, each item is scored from 0-4, total severity score is calculated by taking the sum of the individual item scores (range: 0-80). Higher scores denote greater symptom severity.
  A participant is defined as remitter at any post-baseline timepoint if their CAPS-5 total severity score is less than or equal to 20.
Time Frame: Week 12
Population: Full Analysis Set - All participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | COMP360 Psilocybin
Number analyzed (Participants) | 22
Participants | 12

5. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Total Score From Baseline
Description: SDS is a 5 item scale. The total score is calculated by summing the 3 domains (work/school, social life, and family life - each domain has a 0-10 range). The total score has a range from 0 to 30, with 0 representing no impairment and 30 representing severe impairment.
Time Frame: Week 12
Population: Full Analysis Set - all participants who received study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COMP360 Psilocybin
Number analyzed (Participants) | 21
units on a scale | -14.4 (8.21)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | COMP360 Psilocybin
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COMP360 Psilocybin (N=22)
Visual impairment (Eye disorders) | 3 (3) — Verbatim terms: 1) Visual distortions, mild (eg Crystals in room looking more vibrant), transient, resolved before leaving session, 2) Change in visual perception (patterns, things appear wavy), 3) changes in visual perception (colors moving)
Nausea (Gastrointestinal disorders) | 8 (9)
Crying (General disorders) | 6 (6)
Fatigue (General disorders) | 6 (6)
Chills (General disorders) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Tension headache (Nervous system disorders) | 6 (9)
Headache (Nervous system disorders) | 6 (6)
Paraesthesia (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Hallucination, visual (Psychiatric disorders) | 5 (5)
Euphoric mood (Psychiatric disorders) | 2 (2)
Paranoia (Psychiatric disorders) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (7):
  • Study Protocol: v5.0 (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT05312151/Prot_000.pdf
  • Study Protocol: v4.0 (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT05312151/Prot_001.pdf
  • Study Protocol: v3.0 (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT05312151/Prot_002.pdf
  • Study Protocol: v2.0 (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT05312151/Prot_003.pdf
  • Study Protocol: v1.0 (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT05312151/Prot_004.pdf
  • Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT05312151/SAP_005.pdf
  • Informed Consent Form (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT05312151/ICF_006.pdf